CLINICAL TRIAL: NCT03709290
Title: Cerebrovascular Changes in Multiple Sclerosis Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, safaa omeira ghaly said, Doctor, Assiut University
Other Study IDs: CVSIMSP
Record Dates: First submitted 2018-10-15; First posted 2018-10-17 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1st group: 30 patients were diagnosed with MS according to revised MacDonald's criteria 2017 & collected from Neuropsychiatry department in Assuit university hospital
  Interventions: Radiation: mri
- 2nd group: 30 healthy volunteers subjects matched with age, sex & education level were recruited from outpatient clinic neuropsychiatry department and included only if they had no current or previous history of any neurological illness and their neurological examination was free
  Interventions: Radiation: mri

INTERVENTIONS:
Radiation: mri — mri brain & spinal cord

SUMMARY:
Multiple sclerosis (MS) MS is a chronic disease containing the inflammatory, demyelinating, anddegenerative processes of the central nervous system. The inflammation, microglial activation, astrocyticgliosis, demyelination, and somewhat axonal loss inwhite matter and grey matter was present in the brainsof the patients with MS . Moreover, MS patientspresented a reduction in the cerebral blood flow (CBF)affecting both grey and white matter in positronemission tomography (PET) studies.

MS is the most common autoimmune disorder of the central nervous system. As of 2010, the number of people with MS was 2-2.5 million (approximately 30 per 100,000) globally, with rates varying widely in different regions. MS affects approximately 1000000 people between 17 and 65 years old world wide, the projected prevalence rate of MS for the white US population was 191 per 1000000 and the incidence rate was 7.3 per 1000000 persons .

the contribution of neurodegenerative processes in the disease pathogenesis has been increasingly recognized, especially with respect to possible mechanisms of progression. These may include axonal degeneration, mitochondrial injury, energy failure, hypoxia, oxidative damage, iron accumulation or global cerebral hypoperfusion . Interestingly, Cerebral vasomotor reactivity (CVMR) in MS may be impaired as well.

Although the cause of CVMR impairment in MS is not clear, several potential factors mightcontribute to this phenomenon.

For the purpose of clarity,we divide them into (1) vascular factors, (2) glial factors, and (3)neuronal factors:

1. Vascular factor

   Blood-brain barrier (BBB) disruption might be anotherfactor contributing to CVMR impairment in neurodegenerative disorders. CVMR impairment could also be caused by an increase inthe concentration of vasoconstrictive agents. For instance,endothelin-1 (ET-1) - a potent vasoconstrictor, is overexpressed in the cerebral vessels of MS and elevated in both serumand cerebrospinal fluid of patients with MS.
2. Glial factors

   Reactive astrocytes, i.e. hypertrophied astrocytes that overexpress GFAP (glial fibrillary acidic protein) have been described in virtually all CNS disorders including MS . they could also contribute to CVMR impairment through the production of ET-1 and possibly other vasoconstrictors Another way in which glial cells could contribute to the impairment of CVMR might be associated with their involvement in oxidative stress pathways. Glial pathology may also cause BBB dysfunction.
3. Neuronal factors

It has been shown that cholinergic projections originating from the nucleus basalis induce cerebral vasodilation directly through the release of acetylcholine and indirectly through the stimulation of NO-releasing interneurons . there is evidence of a cholinergic deficit in MS.

From a clinical point of view, reduced white and gray matter CBF in patients with MS has thus far been associated with cognitive manifestations.

Cognitive impairment occurs in 40 to 65% of patients with MS and can have a considerable impact on occupational and social life. also reduced deep gray matter perfusion in MS negatively correlated with fatigue.

Cerebrovascular reactivity (CVR) is an inherent indicator of the dilatory capacity of cerebral arterioles for a vasomotor stimulus for maintaining a spontaneous and instant increase of CBF) in response to neural activation. The integrity of this mechanism is essential to preserving healthy neurovascular coupling. Transcranial Doppler ultrasound (TCD) is defined as a non-invasive ultrasound procedure to evaluate the changes in cerebral blood flow velocity (CBFV) . The high temporal resolution and non-invasive nature of TCD make it a useful tool in the assessment of integrative cerebrovascular function in terms of cerebral reactivity, autoregulation and neurovascular coupling (NVC).

DETAILED DESCRIPTION:
Multiple sclerosis (MS) MS is a chronic disease containing the inflammatory, demyelinating, anddegenerative processes of the central nervous system[FrischerJMet al, 2009]. The inflammation, microglial activation, astrocyticgliosis, demyelination, and somewhat axonal loss inwhite matter and grey matter was present in the brainsof the patients with MS [Wegner C et al, 2006]. Moreover, MS patientspresented a reduction in the cerebral blood flow (CBF)affecting both grey and white matter in positronemission tomography (PET) studies [Sun X et al, 1998].

MS is the most common autoimmune disorder of the central nervous system[Berer K et al,2014]. As of 2010, the number of people with MS was 2-2.5 million (approximately 30 per 100,000) globally, with rates varying widely in different regions. [Milo R et al ,2010] MS affects approximately 1000000 people between 17 and 65 years old world wide, the projected prevalence rate of MS for the white US population was 191 per 1000000 and the incidence rate was 7.3 per 1000000 persons [Mayr WTet al, 2003]. Another study of prevalence of Multiple Sclerosis in Egypt in age group >17years in a population number 21774 was about 13.74 per 100000 [El-Tallawy HNet al, 2013].

The contribution of neurodegenerative processes in the disease pathogenesis has been increasingly recognized, especially with respect to possible mechanisms of progression. These may include axonal degeneration, mitochondrial injury, energy failure, hypoxia, oxidative damage, iron accumulation or global cerebral hypoperfusion [Mahad DH et al, 2015, D'haeseleer M et al, 2015]. Interestingly, Cerebral vasomotor reactivity (CVMR) in MS may be impaired as well.

Although the cause of CVMR impairment in MS is not clear, several potential factors mightcontribute to this phenomenon.

For the purpose of clarity,we divide them into (1) vascular factors, (2) glial factors, and (3) neuronal factors:

1. Vascular factor

   Blood-brain barrier (BBB) disruption might be anotherfactor contributing to CVMR impairment in neurodegenerative disorders [Alvarez JI, et al, 2013]. CVMR impairment could also be caused by an increase inthe concentration of vasoconstrictive agents. For instance,endothelin-1 (ET-1) - a potent vasoconstrictor, is overexpressed in the cerebral vessels of MS and elevated in both serumand cerebrospinal fluid of patients with MS [Haufschild T, et al,2001, D'haeseleer M, et al,2013].
2. Glial factors

   Reactive astrocytes, i.e. hypertrophied astrocytes that overexpress GFAP (glial fibrillary acidic protein) have been described in virtually all CNS disorders including MS [Ben Haim L, et al, 2015]. they could also contribute to CVMR impairment through the production of ET-1 and possibly other vasoconstrictors Another way in which glial cells could contribute to the impairment of CVMR might be associated with their involvement in oxidative stress pathways [Haider L et al, 2011]. Glial pathology may also cause BBB dysfunction [Alvarez JI, et al, 2013].
3. Neuronal factors

It has been shown that cholinergic projections originating from the nucleus basalis induce cerebral vasodilation directly through the release of acetylcholine and indirectly through the stimulation of NO-releasing interneurons [Hamel E. et al, 2006] there is evidence of a cholinergic deficit in MS [Kooi E-J, et al, 2011].

From a clinical point of view, reduced white and gray matter CBF in patients with MS has thus far been associated with cognitive manifestations [-Inglese M, et al, 2008, D'Haeseleer M et al, 2013].

Cognitive impairment occurs in 40 to 65% of patients with MS and can have a considerable impact on occupational and social life [Amato MP, et al, 2001]. also reduced deep gray matter perfusion in MS negatively correlated with fatigue [Vucic S, et al, 2010].

Cerebrovascular reactivity (CVR) is an inherent indicator of the dilatory capacity of cerebral arterioles for a vasomotor stimulus for maintaining a spontaneous and instant increase of CBF) in response to neural activation. The integrity of this mechanism is essential to preserving healthy neurovascular coupling. Transcranial Doppler ultrasound (TCD) is defined as a non-invasive ultrasound procedure to evaluate the changes in cerebral blood flow velocity (CBFV) [Powers J et al,2009]. The high temporal resolution and non-invasive nature of TCD make it a useful tool in the assessment of integrative cerebrovascular function in terms of cerebral reactivity, autoregulation and neurovascular coupling (NVC).

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with MS or diagnosis of CIS highly suggestive of MS according to revised McDonald's criteria 2010.
2. MS patients aged (18-60 years) of both sexes.
3. EDSS score (1-7).

Exclusion Criteria:

1. History or current evidence of CNS diseases other than MS which may affect brain volume &cognition e.g. (Dementia prior to MS, parkinsonism, other inflammatory CNS diseases).
2. History or current evidence of medical illness as endocrinal or metabolic which may affect cognitive function e.g. (hepatic, renal impairment or hypothyrodism).
3. History or current intake of any drug that may affect cognitive function e.g (Antiepileptic, antipsychotic…).
4. History or current evidence of depression (according to DSM -5- criteria &Hamilton depression scale) or any psychiatric disorder.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All patients are subjected to the following:
  1. History taking and full general and neurological examination.
  2. Laboratory tests:
     CBC-KFT-LFT-Na-K-PT-PC-INR..
  3. MRI brain and spinal cord:
     To confirm diagnosis of MS by experienced neuro-radiologist.
  4. Visual Evoked potential:
     Help to confirm diagnosis (detect central demyelination and disseminated in space), VEP was performed using the Nihon Kohden model). MEB-7102 (Nihon Kohden Corp., Tokyo, Japan).
  5. Expanded Disability Status Scale (EDSS) [Kurtzke JF. Et al, 1983]. This scale provides an overall rating of disabilities based on 0(normal neurological examination) to 10 (death due to MS) point scale, higher scores represent greater degree of disability.
  6. Transcranial doppler study
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
evaluate cerebrovascular changes in patients with MS byTCD, which is an easy applicable and non-invasivebedside technique | 1 year

IPD SHARING:
Plan to Share IPD: No